CLINICAL TRIAL: NCT02813772
Title: Efficacy of a Partially Hydrolyzed Formula, Containing Lactobacillus Reuteri, for Infant Colic: a Double Blind, Randomized-controlled Trial
Brief Title: Efficacy of a Partially Hydrolyzed Formula, Containing Lactobacillus Reuteri, for Infant Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annamaria Staiano, Professor of Pediatrics, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30/05/2016
Record Dates: First submitted 2016-06-14; First posted 2016-06-27 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Infant Colics
Keywords: infants; colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Experimental): Patients with infantile colics who will receive the milk formula NAN Sensitive, Nestlè
  Interventions: Dietary Supplement: Milk formula NAN Sensitive, Nestle
- group 2 (Active Comparator): Patients with infantile colics who will receive the milk formula NAN Optipro, Nestlè
  Interventions: Dietary Supplement: Milk formula Optipro, Nestle

INTERVENTIONS:
Dietary Supplement: Milk formula NAN Sensitive, Nestle — Infants randomized to group 1 will receive the milk formula NAN Sensitive, Nestle for a period of 4 weeks.
  Arms: group 1
Dietary Supplement: Milk formula Optipro, Nestle — Infants randomized to group 1 will receive the milk formula NAN Optipro, Nestle for a period of 4 weeks.
  Arms: group 2

SUMMARY:
Infant colic (IC) is responsible of 25% of pediatric consultation in the first 3-4 months of life affecting from 5% to 30% of infants between 2 weeks and 3 months of life (3, 4). The variability in the prevalence of IC reported by the several studies depends on different criteria used to define IC.The etiology of IC remains still unclear. Recently, the composition of intestinal microbiome has been addressed as an independent risk factor for IC. There are no uniform criteria for a specific therapeutic approach of IC. Based on these conclusions the objectives of our study are: to determine whether the administration of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri, is beneficial in IC in reducing the infant crying duration and in prolonging the duration of sleeping period

DETAILED DESCRIPTION:
BACKGROUND Definition Infantile Colic (IC) is one of the Functional gastrointestinal disorders (FGIDs) of infants/toddlers, which are defined as a variable combination of chronic or recurrent gastrointestinal symptoms not explained by structural or biochemical abnormalities. In 2006, the Rome III committee established a new criteria defining it as "episodes of irritability, fussing, or crying that begin and end for no apparent reason and last at least three hours a day, at least three days a week, for at least one week".

Epidemiology IC is responsible of 25% of pediatric consultation in the first 3-4 months of life affecting from 5% to 30% of infants between 2 weeks and 3 months of life. The variability in the prevalence of IC reported by the several studies depends on different criteria used to define IC.

In a systematic review of 15 community-based surveys on IC prevalence, carried out in 2001, the occurrence rates in the first 3 months of life were from 3% to 28% in prospective studies and from 8% and 40% in retrospective studies. In a prospective study found that 20.5% of 2879 Italian infants, aged 2 weeks-6 months, had IC.

Recently a French study reported a prevalence of IC in infants aged 0-4 months, of 19%. In two english studies, IC was reported in 18.3% and 26 % respectively, of infants aged 0-12 months. Other European studies were conducted with a different reported prevalence.

Outside Europe, a prevalence of 9.2% and of 20% respectively were reported by two studies carried out in US. More recently in an Israeli study of 94 mothers of 2-4 moths of life infants, 56% of those whose babies were breastfed and 73% of those using formula reported "paroxysmal irritability".

In addition, several studies found occurrence rates of crying/fussing problems in young infants ranging from 7% to 19%, without defining the problems as IC.

Pathogenesis The etiology of IC remains still unclear. Gender, type of milk (breast-milk or formula), delivery modality (vaginally or caesarean), mother age, number of siblings and gestational history do not seem to be correlated to IC onset. Gastrointestinal function, psychosocial, and neurodevelopmental disorders, food intolerance, transient low lactase activity, cow's milk protein allergy (CMPA), gastro-esophageal reflux (GER) and intestinal microbiota imbalance have been suggested as the cause of colic.

Gastrointestinal theories include increased intra-abdominal gas, hyperperistalsis and visceral pain. Gastrointestinal disorders have been implicated in colic because of the infant's leg position and grimacing during the crying episodes. Excessive crying or increased gas production from colon function can result in intraluminal gas formation and aerophagia, even if radiographic images taken during a crying episode have shown a normal gastric outline. One study has suggested that infants with colic may have increased fecal calprotectin levels, suggesting a possible role for gut inflammation; however, another study suggested no differences in fecal calprotectin levels between infants with and infants without colic. Gut hormones, such as motilin, also may play a causative role in colic. Motilin is thought to cause hyperperistalsis, leading to abdominal pain and colic. Regarding psychosocial hypotheses, maternal anxiety and depression, and difficult infant temperament have been correlated to IC. Also behavioral issues such as family tension or inadequate interaction between parents and infant have been considered, but these issues are really controversial. Concomitant risk factors remain partially unknown; however, maternal smoking, increased maternal age and firstborn status may be associated to the development of IC.

The role of intestinal microbiome in Infantile Colic Recently, the composition of intestinal microbiome has been addressed as an independent risk factor for IC. Several studies indicate that inadequate lactobacilli in the first few months of life may affect intestinal fatty acid profile favoring the development of IC. Coliform bacteria have also been found more abundantly in colicky infants and it is speculated that altering the intestinal microbiota composition may positively influence the management of affected infants. As a matter of fact, recently, research into the use of probiotics for colic has been rapidly increasing but results are conflicting. Infants with colic are reported to have increased concentration of gas forming organisms and proteobacteria such as Escherichia coli in their gut. Colonization with certain intestinal microorganisms, such as Bifidobacterium and Lactobacillus species, along with increased intestinal microbial diversity, may protect against infant distress. Probiotics enhance the mucosal barrier and promote microbial diversity in the gut. They may reduce concentrations of proteobacteria and gas forming coliform and reduce intestinal inflammation.

One clinical trial showed safety and efficacy of Lactobacillus reuteri in prevention of IC. A recent meta-analysis of three small, randomized controlled trials, of breast-fed infants with IC reported that Lactobacillus reuteri noticeably reduced crying time at 21 days post supplementation. Recently Chau et al showed that administration of Lactobacillus reuteri DSM 17938 significantly improved colic symptoms by reducing crying and fussing times in breastfed Canadian infants with colic. In contrast, a double blind, placebo controlled randomized trial on the same probiotic strain Lactobacillus reuteri DSM 17938 showed that it did not benefit a community sample of breast-fed infants and formula-fed infants with IC.

The role of diet in Infant colic There are no uniform criteria for a specific therapeutic approach of IC. Regarding dietary modifications on management of IC, current evidence suggests that they may reduce IC in only a very small minority of infants. Unfortunately, the evidence is often contrasting. For the breast-fed infants with IC, where there is the relatively rare concern of a cow's milk protein allergy (CMPA), one can consider eliminating cow's milk from the maternal diet for a minimum of two weeks. For the formula-fed infants with colic, the use of a time-limited (two weeks) empiric trial of an extensively hydrolyzed formula may be considered. However this information derived from studies in highly selected patients from tertiary care level centers. In a double-blind, placebo-controlled trial, a partial hydrolyzed, with high β-palmitate, and a specific prebiotics mixture with galacto- and fructo-oligosaccharides resulted in a significant decrease of colic within one week of intervention. In some cases, these formulas are lactose-reduced or lactose-free and contain prebiotics or probiotics causing a reduction in the number of crying episodes per week and total crying time. Infante et al showed an association between clinical improvement and evidence of decreased levels of hydrogen in IC when the infants were fed with a specially designed, low-lactose formula. Moreover, in two double-blinded crossover trials, lactase treatment reduced crying time compared with placebo. The use of soy formulas, instead, in the treatment of IC should be avoided since it can induce sensitization to soy and it's high in isoflavones with estradiol-like effects.

OBJECTIVES

Primary objective:

-To determine whether the administration of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri, is beneficial in IC in reducing the infant crying duration.

Secondary objectives:

* To evaluate the effect of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri in prolonging the duration of sleeping period.
* To evaluate the effect of this infant formula enriched with Lactobacillus reuteri on fecal microbiome of colicky infants
* To evaluate the effect of this infant formula enriched with Lactobacillus reuteri on parents' quality of life
* To evaluate the effect of this infant formula enriched with Lactobacillus reuteri on infants' quality of life

METHODS

Study design

* This is a prospective, double-blind, randomized-controlled, clinical trial.
* The study aims to compare the infant colic's trend and intestinal microbiome between infants fed with partially hydrolyzed formulas (pHF; 100% whey protein; 1.9g/100 kcal) with reduced lactose content (40%), addition of maltodextrins (60%) and Lactobacillus reuteri (NAN Sensitive, Nestlè) (group 1) and infants fed with an intact protein body formula (70% of whey protein, 30% of casein; 1.85g/100 kcal) with 100% of lactose content and not containing Lactobacillus reuteri (NAN Optipro 1, Nestlè) (group 2).
* Subjects will be enrolled consecutively and randomized to one of the 2 study groups.

ELIGIBILITY:
Inclusion Criteria:

Full-term infants (≥37 weeks gestation at birth); Exclusively formula fed infants at time of enrolment; Infants suffering from IC according to Rome III criteria (Appendix 1); Age < 4 months of life; 5-minute Apgar score ≥7; Birth weight ≥2500 g.

Exclusion Criteria:

Consumption of formula containing probiotics, pHF or with reduced lactose content at time of enrolment; Major medical problem or acute illness, including gastroesophageal reflux, cow's milk protein allergy History of antibiotic treatment before or during the study; History of probiotic or L reuteri supplementation; History of any allergies to any of the ingredients in the probiotic L reuteri Concurrent participation in another clinical trial. Birth weight < 2500 g; Failed to thrive; Breastfed infants; NAN (to avoid the formula switch effect).

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
whether the administration of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri, is beneficial in IC in reducing the infant crying duration. | 7, 14, 21, 28 days, 2 and 3 months
  Infant crying duration (minutes per day) at 7, 14, 21, 28 days, 2 and 3 months post-intervention.

SECONDARY OUTCOMES:
whether the administration of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri, is beneficial in IC in reducing the infant crying duration. | 28 days
  Percentage of responders at 28 days post-intervention. A response to the treatment will be defined as 50% of reduction of infant crying.
whether the administration of a partially hydrolyzed formula (pHF) with reduced lactose content and Lactobacillus reuteri, is beneficial in IC in increasing infant sleep. | 7, 14, 21, 28 days, 2 and 3 months
  Longer infant sleep duration at 7, 14, 21, 28 days, 2 and 3 months post-intervention
the effect of a partially hydrolyzed formula (pHF) on quality of life of the enrolled patients | 3 months
  Reduction of mean scores of a standardized measure for childrens' quality of life
the effect of a partially hydrolyzed formula (pHF) on quality of life of parents | 3 months
  Reduction of mean scores of a standardized measure for parents' quality of life
the effect of this infant formula enriched with Lactobacillus reuteri on fecal microbiome of colicky infants | 2 months
  Changes in gut microbiome
Changes in stool frequency and consistency | 28 days
  Changes in stool frequency and consistency
Parental perception of colic severity (VAS 0-10) | 28 days
  Parental perception of colic severity (VAS 0-10)
Parental perception of sleep quality (VAS 0-10) | 28 days
  Parental perception of sleep quality (VAS 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Annamaria Staiano, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
December 2016

REFERENCES:
- [Derived] Turco R, Russo M, Bruzzese D, Staiano A. Efficacy of a partially hydrolysed formula, with reduced lactose content and with Lactobacillus reuteri DSM 17938 in infant colic: A double blind, randomised clinical trial. Clin Nutr. 2021 Feb;40(2):412-419. doi: 10.1016/j.clnu.2020.05.048. Epub 2020 Jun 12. PMID 32600858